CLINICAL TRIAL: NCT01595126
Title: A Longitudinal Study of Biomarkers in Pediatric Patients With Central Nervous System Tumors
Brief Title: Longitudinal Study of Biomarkers
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-14877
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Central Nervous System Tumor
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Central Nervous System Tumors

SUMMARY:
Biomarkers are small molecules that can be detected in the body fluids of patients; they often correlate with the presence of a cancer. MicroRNAs and proteins are small molecules which have recently been discovered in cells. They are known to be responsible for the normal development of cells and when they are disrupted can contribute to the development of cancer. Many previous studies have been done evaluating the expression of microRNAs and proteins in normal tissues as well as a wide variety of cancers.

Recently, microRNAs and proteins from tumor cells have been detected circulating in the blood of patients with cancer. This presents a novel opportunity to use microRNAs and proteins in the blood as an early predictor of cancer as well as a marker of response to therapy. Previous work in our labs have identified miRNAs and proteins in the blood and cerebrospinal fluid (CSF) of pediatric patients with brain tumors.

To determine a longitudinal evaluation of the presence of microRNAs and proteins in the blood, cerebrospinal fluid and urine of patients with central nervous system tumors from diagnosis through the course of their treatment. Though the duration of active treatment varies significantly based upon the diagnosis, patients will be followed for up to 24 months after enrollment onto the study).

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 1 day to 21 years
* Patients with radiographically and/or histologically confirmed CNS tumors treated at Children's Memorial Hospital and Lurie Children's Hospital in Chicago
* Patients must be newly diagnosed and have had no prior anticancer therapy (except surgery) for their current diagnosis. The use of steroids is permissible.
* Patients and/or parents/legal guardians must have signed an informed consent and assent when applicable.

Exclusion Criteria:

* Patients who have completed treatment and do not require routine blood draws and/or lumbar punctures
* Patients who are considered too ill to participate as determined by their treating physician
* Patients who are pregnant or lactating

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly diagnosed patients with central nervous system tumors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Presence of microRNAs and proteins in the blood, cerebrospinal fluid and urine of patients with central nervous system tumors from diagnosis through the course of their treatment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Lulla, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Fernandez-L A, Northcott PA, Taylor MD, Kenney AM. Normal and oncogenic roles for microRNAs in the developing brain. Cell Cycle. 2009 Dec 15;8(24):4049-54. doi: 10.4161/cc.8.24.10243. Epub 2009 Dec 5. PMID 19901543
- [Background] Birks DK, Barton VN, Donson AM, Handler MH, Vibhakar R, Foreman NK. Survey of MicroRNA expression in pediatric brain tumors. Pediatr Blood Cancer. 2011 Feb;56(2):211-6. doi: 10.1002/pbc.22723. Epub 2010 Nov 3. PMID 21157891
- [Background] Sredni ST, Huang CC, Bonaldo Mde F, Tomita T. MicroRNA expression profiling for molecular classification of pediatric brain tumors. Pediatr Blood Cancer. 2011 Jul 15;57(1):183-4. doi: 10.1002/pbc.23105. Epub 2011 Mar 21. No abstract available. PMID 21425446
- [Background] Taylor DD, Gercel-Taylor C. MicroRNA signatures of tumor-derived exosomes as diagnostic biomarkers of ovarian cancer. Gynecol Oncol. 2008 Jul;110(1):13-21. doi: 10.1016/j.ygyno.2008.04.033. PMID 18589210
- [Background] Lawrie CH, Gal S, Dunlop HM, Pushkaran B, Liggins AP, Pulford K, Banham AH, Pezzella F, Boultwood J, Wainscoat JS, Hatton CS, Harris AL. Detection of elevated levels of tumour-associated microRNAs in serum of patients with diffuse large B-cell lymphoma. Br J Haematol. 2008 May;141(5):672-5. doi: 10.1111/j.1365-2141.2008.07077.x. Epub 2008 Mar 3. PMID 18318758
- [Background] Huang Z, Huang D, Ni S, Peng Z, Sheng W, Du X. Plasma microRNAs are promising novel biomarkers for early detection of colorectal cancer. Int J Cancer. 2010 Jul 1;127(1):118-26. doi: 10.1002/ijc.25007. PMID 19876917
- [Background] Ng EK, Chong WW, Jin H, Lam EK, Shin VY, Yu J, Poon TC, Ng SS, Sung JJ. Differential expression of microRNAs in plasma of patients with colorectal cancer: a potential marker for colorectal cancer screening. Gut. 2009 Oct;58(10):1375-81. doi: 10.1136/gut.2008.167817. Epub 2009 Feb 6. PMID 19201770
- [Background] Ji X, Takahashi R, Hiura Y, Hirokawa G, Fukushima Y, Iwai N. Plasma miR-208 as a biomarker of myocardial injury. Clin Chem. 2009 Nov;55(11):1944-9. doi: 10.1373/clinchem.2009.125310. Epub 2009 Aug 20. PMID 19696117
- [Background] Ai J, Zhang R, Li Y, Pu J, Lu Y, Jiao J, Li K, Yu B, Li Z, Wang R, Wang L, Li Q, Wang N, Shan H, Li Z, Yang B. Circulating microRNA-1 as a potential novel biomarker for acute myocardial infarction. Biochem Biophys Res Commun. 2010 Jan 1;391(1):73-7. doi: 10.1016/j.bbrc.2009.11.005. Epub 2009 Nov 5. PMID 19896465
- [Background] Das T, Bae YH, Wells A, Roy P. Profilin-1 overexpression upregulates PTEN and suppresses AKT activation in breast cancer cells. J Cell Physiol. 2009 Feb;218(2):436-43. doi: 10.1002/jcp.21618. PMID 18937284
- [Background] Kolwijck E, Kos J, Obermajer N, Span PN, Thomas CM, Massuger LF, Sweep FC. The balance between extracellular cathepsins and cystatin C is of importance for ovarian cancer. Eur J Clin Invest. 2010 Jul;40(7):591-9. doi: 10.1111/j.1365-2362.2010.02305.x. Epub 2010 May 12. PMID 20482593
- [Background] Srikantha U, Balasubramaniam A, Santosh V, Somanna S, Bhagavatula ID, Ashwathnarayana CB. Recurrence in medulloblastoma - influence of clinical, histological and immunohistochemical factors. Br J Neurosurg. 2010 Jun;24(3):280-8. doi: 10.3109/02688691003660558. PMID 20465457
- [Background] Smyth GK. Linear models and empirical bayes methods for assessing differential expression in microarray experiments. Stat Appl Genet Mol Biol. 2004;3:Article3. doi: 10.2202/1544-6115.1027. Epub 2004 Feb 12. PMID 16646809
- [Background] Liu H, Sadygov RG, Yates JR 3rd. A model for random sampling and estimation of relative protein abundance in shotgun proteomics. Anal Chem. 2004 Jul 15;76(14):4193-201. doi: 10.1021/ac0498563. PMID 15253663